CLINICAL TRIAL: NCT04420611
Title: Use of Endogenous Melatonin and 6-hydroxymelatonin as Biomarkers for CYP1A2
Acronym: MelaCYP
Status: Completed | Type: Observational
Sponsor: Youssef Daali (Other)
Responsible Party: Sponsor-Investigator, Youssef Daali, Professor Youssef Daali, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: 2020-00125
Record Dates: First submitted 2020-05-19; First posted 2020-06-09 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * 12-hour urine collection during the night (21h-9h) with the first urine in the morning collected separately
  * capillary blood samples (10 μL)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Session 1 (day 1) — 12 hours overnight urine (9 pm - 9 am) will be collected. First morning voids will be collected separately in order to be also analysed independently from the 12 hours collection. 24 hours before the 12 hours overnight urine collection, volunteers will be asked to refrain from alcohol consumption and methylxanthine-containing beverages and foods.
  After the 12-hour urine collection (around 9:00 a.m.), subjects will be given a cup of coffee or a can of Coca-Cola®. Capillary blood samples (10 μL) will be taken from the fingertips 2 hours after the coffee or Coca-Cola®.
Other: Session 2 (day 3) — 12 hours overnight urine (9 pm - 9 am) will be collected. First morning voids will be collected separately in order to be also analysed independently from the 12 hours collection. 24 hours before the 12 hours overnight urine collection, volunteers will be asked to refrain from alcohol consumption and methylxanthine-containing beverages and foods.
  After the 12-hour urine collection (around 9:00 a.m.), subjects will be given a cup of coffee or a can of Coca-Cola®. Capillary blood samples (10 μL) will be taken from the fingertips 2 hours after the coffee or Coca-Cola®.
Other: Session 3 (day 15) — 12 hours overnight urine (9 pm - 9 am) will be collected. First morning voids will be collected separately in order to be also analysed independently from the 12 hours collection. 24 hours before the 12 hours overnight urine collection, volunteers will be asked to drink or eat caffeinated food/drinks 24 hours prior to night-time urine collection (at least one cup of coffee or a can of Coca-Cola®).
  After the 12-hour urine collection (around 9:00 a.m.), subjects will be given a cup of coffee or a can of Coca-Cola®. Capillary blood samples (10 μL) will be taken from the fingertips 2 hours after the coffee or Coca-Cola®.
Other: Session 4 (day 30) — 12 hours overnight urine (9 pm - 9 am) will be collected. First morning voids will be collected separately in order to be also analysed independently from the 12 hours collection. 24 hours before the 12 hours overnight urine collection, volunteers will be asked to refrain from alcohol consumption and methylxanthine-containing beverages and foods.
  After the 12-hour urine collection (around 9:00 a.m.), subjects will be given a cup of coffee or a can of Coca-Cola®. Capillary blood samples (10 μL) will be taken from the fingertips 2 hours after the coffee or Coca-Cola®.

SUMMARY:
An observational study comprising 4 sessions will be conducted in 12 healthy volunteers. During each study session (sessions 1 to 4), a 12-hour urine collection during the night (21h-9h) will be carried out by each participant. The first urine in the morning will be collected separately to be analysed independently of the 12-hour collection. 24 hours before the start of the night urine collection, volunteers will be asked to refrain from consuming alcohol and caffeinated drinks/foods, with the exception of session 3. Conversely, in session 3, subjects will be asked to drink or eat caffeinated food/drinks 24 hours prior to night-time urine collection (at least one cup of coffee or a can of Coca-Cola®).

After each 12-hour urine collection (around 9:00 a.m.), subjects will be given a cup of coffee or a can of Coca-Cola®. Capillary blood samples (10 μL) will be taken from the fingertips 2 hours after the coffee or Coca-Cola®.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Understanding of French language and ability to give a written informed consent

Exclusion Criteria:

* Inability to refrain from alcohol or methylxanthine-containing beverages and foods for 24 hours
* Sensitivity to coffee or CocaCola®
* Irregular (i.e. non-daily or inconstant dosages) intake of medication or food of a CYP1A2 modulator (including tobacco)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy men and women
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Validation LC-MS/MS analytical method | 1 month
  Validation of the LC-MS/MS analytical method for simultaneous quantification of endogenous melatonin and 6-hydroxymelatonin in urine samples

SECONDARY OUTCOMES:
Intra- and inter-variability | 3 days (day 1, day 4 and day 30)
  Assess intra- and inter-variability of the urinary metabolic ratio (UMR) 6-hydroxymelatonin/melatonin at three different time (day 1, day 4 and day 30)
Urine correlation | 4 days (day 1, day 4, day 15 and day 30)
  Assess correlation between 12 hours overnight urine and first morning voids samples
Correlation melatonin and caffeine | 4 days (day 1, day 4, day 15 and day 30)
  Assess correlation between the endogenous UMR 6-hydroxymelatonin/melatonin and the paraxanthine/caffeine ratio in dried blood spot (DBS)
Impact caffeine intake | 1 day (day 15)
  Assess impact of caffeine intake on the UMR 6-hydroxymelatonin/melatonin (day 15) before and after caffeine abstinence (fold-change measurements)

CONTACTS AND LOCATIONS:
Overall Officials: Youssef Daali, Prof, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland